CLINICAL TRIAL: NCT07247643
Title: The Impact of Virtual Reality Glasses on Maternal Satisfaction and Postpartum Comfort in Cesarean Sections Performed Under Spinal Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Büşra Küçüktürkmen (Other)
Responsible Party: Sponsor-Investigator, Büşra Küçüktürkmen, Research Assistant, Department of Midwifery, Bilecik Seyh Edebali Universitesi
Organization: Bilecik Seyh Edebali Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-10333602-050.04-280407
Record Dates: First submitted 2025-09-07; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Caesarean Section
Keywords: caesarean section; virtual reality; cesarean birth satisfaction; postpartum comfort; spinal anesthesia
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Intervention Group): Virtual Reality Glasses (Experimental): Participants in this group will undergo cesarean section under spinal anesthesia and, during the procedure, will watch immersive nature videos with sound through virtual reality (VR) glasses. The VR application will be paused at the time of birth to allow for initial newborn care and skin-to-skin contact, and then resumed until the completion of suturing. In addition to the VR application, all participants will also receive standard perioperative care that is routinely provided to patients undergoing cesarean delivery.
  Interventions: Device: (Intervention Group): Virtual Reality Glasses
- Control Group (Other): Participants in this group will undergo cesarean section under spinal anesthesia and will receive routine perioperative care only, without the use of virtual reality.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: (Intervention Group): Virtual Reality Glasses — Participants in this group will undergo cesarean section under spinal anesthesia and, during the procedure, will watch immersive nature videos with sound through virtual reality (VR) glasses. The VR application will be paused at the time of birth to allow for initial newborn care and skin-to-skin contact, and then resumed until the completion of suturing. Standard perioperative care will also be provided.
  Arms: (Intervention Group): Virtual Reality Glasses
Other: Control Group — Participants in this group will undergo cesarean section under spinal anesthesia and will receive routine perioperative care only, without the use of virtual reality.
  Arms: Control Group

SUMMARY:
Due to the stressful nature of cesarean birth, it is important that the use of virtual reality (VR) glasses is both feasible and effective. While wearing VR glasses, the distraction effect can reduce women's focus on pain and the surgical procedure itself. Furthermore, VR applications have been shown to increase women's satisfaction with the birth experience. This study will be conducted as a randomized controlled trial. A total of 96 participants will be included, with 48 assigned to the intervention group and 48 to the control group. The intervention group will consist of women undergoing repeat cesarean section under spinal anesthesia. During the procedure, participants in the intervention group will watch nature videos with sound through VR glasses. The VR application will be paused when the baby is born to allow for initial neonatal care and skin-to-skin contact. After skin-to-skin contact has been established, the VR application will resume and continue until the completion of the suturing process. Subsequently, once the women are transferred to the ward, the "Personal Information Form," the "Postpartum Comfort Scale," and the "Cesarean Birth Satisfaction Scale for Women Under Spinal Anesthesia," developed by the researcher, will be administered at an appropriate time. This study is expected to support healthcare professionals in integrating VR technology into childbirth practices by providing insights into women's experiences with this intervention. In this way, the study aims to reduce negative emotions experienced during cesarean birth, support the postpartum recovery process, and enhance overall patient satisfaction. Moreover, the findings will contribute to improving the feasibility of digital innovations in healthcare, enhancing the quality of birth experiences, and strengthening the approach to patient-centered care.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18-45 years

Undergoing elective repeat cesarean section under spinal anesthesia

Able to communicate in Turkish and provide informed consent

Singleton pregnancy

Exclusion Criteria:

Presence of obstetric or medical complications requiring general anesthesia

Emergency cesarean sections

Psychiatric or neurological disorders that may interfere with VR use

Contraindications to spinal anesthesia

Visual or hearing impairments preventing effective use of VR glasses

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Cesarean Birth Satisfaction | Within 48 hours after cesarean delivery
  Women's satisfaction with their cesarean delivery experience will be assessed using the researcher-developed "Cesarean Delivery Satisfaction Scale for Women Under Spinal Anesthesia." It will be measured using a researcher-developed 11-item, 5-point Likert-type scale (scores range from 11 to 55), with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Postpartum Comfort | Within 48 hours after cesarean delivery
  Women's postpartum comfort will be measured using the "Postpartum Comfort Scale." It uses a 5-point Likert-type scoring system. The lowest possible score is 34, and the highest is 170. Higher scores indicate greater comfort.